CLINICAL TRIAL: NCT03826563
Title: Melatonin Effects on Sleep and Circadian Rhythm in Youth and Young Adults With At-risk Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: University of Pennsylvania (Other); Brain and Behavior Research Foundation (NARSAD Young Investigator Award, Grant Number 26742) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 18-014932
Record Dates: First submitted 2019-01-17; First posted 2019-02-01 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Psychosis; Sleep
MeSH Terms: conditions — Psychotic Disorders | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Only the pharmacy will know the randomization arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Subjects will receive pill placebo nightly
  Interventions: Other: Placebo
- Melatonin (Experimental): Subjects will receive oral melatonin tablets 2.5-10mg nightly for 2 weeks. All will receive melatonin 5mg for one week, then at the 1 week visit, the dose can be continued at 5mg or adjusted to 2.5mg or 10mg nightly based on clinical assessment of patient response and side effects.
  Interventions: Drug: oral melatonin tablets (NatureMade brand)

INTERVENTIONS:
Drug: oral melatonin tablets (NatureMade brand) — melatonin tablets
  Arms: Melatonin
Other: Placebo — pill placebo
  Arms: Placebo

SUMMARY:
Randomized control trial assessing supplemental melatonin for youth with at-risk or psychotic symptoms.

DETAILED DESCRIPTION:
Context: Sleep disturbances and circadian dysrhythmias have been associated with psychotic symptom severity in Psychosis Spectrum (PS) youths. Supplemental melatonin is a safe over-the-counter dietary supplement, and several studies have found that melatonin improves sleep across several childhood neuropsychiatric disorders.

Objectives: Investigators seeks to determine whether supplemental melatonin improves sleep and circadian alignment in PS youth. Investigators will also investigate whether supplemental melatonin affects psychotic symptoms, neurocognition, and peripheral inflammatory and oxidative stress markers.

Study Design: Parallel group, double-blind, randomized, placebo-controlled trial Setting/Participants: 40 PS youths ages 11-30 years old (throughout the protocol we use "youth" to describe this age group) with sleep disturbances will be recruited from an extant cohort of PS youths followed by our lab in the Philadelphia Neurodevelopmental Cohort (PNC), Children's Hospital of Philadelphia (CHOP), University of Pennsylvania (UPenn), and the surrounding community. The study will be conducted at CHOP and UPenn.

Study Interventions and Measures: Youths will be randomized to receive pill placebo or oral melatonin. Participants will take melatonin (or placebo) at the same time every evening for 2 weeks (final dose range 2.5-10 mg nightly). Outcomes will be assessed at 1 week, 2 weeks, and 6-months. Primary outcomes will be changes in self-reported sleep and actigraph-measured sleep and circadian rhythm. Secondary outcomes will be psychotic symptoms, neurocognition, and peripheral blood markers of inflammation and oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

* Males or females age 11-30 years old and patient at the Children's Hospital of Philadelphia (CHOP), University of Pennsylvania (UPenn), or member of the surrounding community
* Subthreshold psychosis-risk positive symptoms (e.g. hallucinations or unusual beliefs) on the Structured Interview of Psychosis-Risk Syndromes (SIPS)
* At least mild sleep disturbances on the SIPS (>=1 on the SIPS sleep item (G1)) with difficulties with
* Must have difficulties with sleep onset, sleep awakenings, or maintaining a regular sleep schedule.
* Willingness to report all changes in medications and therapy during the study
* Intelligence Quotient (IQ) > 70
* If female, not breastfeeding and not pregnant and willing to use effective birth control for the duration of the study (e.g. abstinence or oral contraception).
* Medically healthy
* Fluent in English

Exclusion Criteria:

* Psychiatric symptoms with imminent safety concern (e.g. intractable and escalating suicidal ideation)
* Currently taking melatonin, having taken melatonin daily within the 2 weeks prior to Visit 1, or having a history of an intolerance or allergy to melatonin.
* Medication or treatment changes in the 4 weeks prior to Visit 1 .
* Anticipated medication or other treatment (e.g. type of psychotherapy) changes in the three weeks after study enrollment.
* IQ <70
* Taking any medication whose potential interactions with melatonin present a significant risk or limit the effect of melatonin in the judgment of the investigators.

Ages: 11 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2023-04-07 (Actual); Study Completion 2023-04-07 (Actual)

PRIMARY OUTCOMES:
Actigraph-measured sleep (increased total sleep time) | Change in total sleep time from melatonin randomization day (Day 0) to Day 14
  Actigraph-measured total sleep time will be used to assess actigraph-measured sleep efficacy, Actigraphs from the Actigraph Company will be used to analyze the data using Actilife software.

SECONDARY OUTCOMES:
Improved self-reported sleep | Change in total PSQI from melatonin randomization day (Day 0) to Day 14
  Pittsburgh Sleep Quality Index (PSQI); range is 0-21, with higher scores indicating poorer sleep

OTHER OUTCOMES:
Decreased actigraph-measured sleep latency | Change in actigraph-measured sleep onset latency from melatonin randomization day (Day 0) to Day 14
  How long it takes a participant to fall asleep; Actigraphs from the Actigraph Company will be used to analyze the data using Actilife software. Sleep latency is an Actilife software outcome.
Increased actigraph-measured sleep efficiency | Change from Randomization day (Day 0) to Day 14.
  Amount of time participant spends sleeping divided by the amount of time the patient spends in bed. Actigraphs from the Actigraph Company will be used to analyze the data using Actilife software. Sleep efficiency is an Actilife software outcome.
Lower autocorrelation function | Change in actigraph-measured autocorrelation from melatonin randomization day (Day 0) to Day 14
  Ac is the slope of the time correlation line (log-trans- formed); indicative of rhythm fragmentation; lower values represent less fragmented rhythms. Actigraphs from the Actigraph Company will be used to analyze the data using Actilife software. Autocorrelation function is an Actilife software outcome.
Increased activity (M10) | Change in actigraph-measured M10 from melatonin randomization day (Day 0) to Day 14
  mean activity level during the most active 10 h of the day; higher values are indicative of a more active lifestyle. M10 is an Actilife software output.

CONTACTS AND LOCATIONS:
Overall Officials: Raquel Gur, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
We will share data within the CHOP research group.